CLINICAL TRIAL: NCT02171897
Title: Comparison of Functional Recovery After Pertrochanter Fracture Treated With Either Total Hip Replacement or Centromedullary Nailing
Brief Title: Pertrochanter Arthroplasty Versus Osteosynthesis
Acronym: PAVO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: TREMLET AOI 2013
Record Dates: First submitted 2014-06-18; First posted 2014-06-24 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Pertrochanter Fracture
MeSH Terms: interventions — Fracture Fixation, Internal; Arthroplasty, Replacement, Hip

ARMS (2):
- Patients treated with osteosynthesis (Experimental)
  Interventions: Procedure: Osteosynthesis
- Patients treated with total hip replacement (Experimental)
  Interventions: Procedure: Total hip replacement

INTERVENTIONS:
Procedure: Osteosynthesis
  Arms: Patients treated with osteosynthesis
Procedure: Total hip replacement
  Arms: Patients treated with total hip replacement

SUMMARY:
This is a single-centre, comparative, prospective randomised trial. It will include 70 patients over a period of 2 years randomized into two groups of 35 patients: one group of patients treated with osteosynthesis (plate, nail or screw) and the second group treated with total hip replacement.

The Harris and PMA functional scores will be assessed at 6 weeks, 3 months, 6 months and 1 year.

The time to recovery of weight-bearing, the subjective satisfaction score, the EQ5D quality of life questionnaire, the VAS score for pain at rest and when walking, the Parker score, the rate of complications and deaths will also be measured. Operating time, blood loss and scar size will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have provided written informed consent
* Patients over 18 years old
* Patients less than 70 years old
* Patient presenting with a fracture of the trochanter (type 1 to 6 according to the Ender classification, and A1 and A2 according tyo the AO classification (Association suisse pour l'étude de l'Ostéosynthèse : classification internationale)

Exclusion Criteria:

* Adult under guardianship
* Patients not covered by national health insurance
* Pregnant or breast-feeding women
* Unable to walk independently before the trauma
* Patients with dementia

Min Age: 70 Years | Sex: All
Age Groups: Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-01-29 (Actual); Primary Completion 2018-10-21 (Actual); Study Completion 2018-10-21 (Actual)

PRIMARY OUTCOMES:
Harris Score | At 6 months after surgery
  Functional hip score

SECONDARY OUTCOMES:
PMA functional score | Up to 1 year after surgery
  Functional score
Time to recovery of weight-bearing | Up to 1 year after surgery
Subjective satisfaction score (EQ5D, VAS score for pain at rest and when walking) | Up to 1 year after surgery
Parker score | Up to 1 year after surgery
  Score autonomy
Rate of complications (loosening of implants, fractures around osteosynthesis devices or prostheses, infections, phlebitis-pulmonary embolism) | Up to 1 year after surgery
Death rate | Up to 1 year after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de DIJON, Dijon, France